CLINICAL TRIAL: NCT00004554
Title: Sertraline for Alcohol Dependence and Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAPET09544
Record Dates: First submitted 2000-02-04; First posted 2000-02-07 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2013-09

CONDITIONS: Alcoholism; Depression
MeSH Terms: conditions — Alcoholism; Depression | interventions — Naltrexone; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sertraline (Experimental): sertraline
  Interventions: Drug: sertraline (Zoloft)
- Naltrexone (Experimental): naltrexone
  Interventions: Drug: naltrexone (Revia)
- Nal/Sert (Experimental): naltrexone/sertraline
  Interventions: Drug: naltrexone (Revia); Drug: sertraline (Zoloft)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: naltrexone (Revia) — 100mg/day
  Arms: Nal/Sert; Naltrexone
Drug: sertraline (Zoloft) — 200mg/day
  Arms: Nal/Sert; Sertraline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will examine depressed alcoholic outpatients to assess whether combining naltrexone (Revia) and sertraline (Zoloft) will result in greater reductions in both drinking and depression over either medication alone or placebo. A secondary aim is to determine whether certain patient features will predict response to sertraline, naltrexone or the combination of the two drugs. Subjects will be randomized into treatment groups for 14 weeks. The followup phase includes two visits at 6 and 9 months after treatment.

DETAILED DESCRIPTION:
The proposed study will examine managing relapse in patients with alcohol dependence and depression using a 14-week double-blind, placebo-controlled, combination of 100 mg/day of naltrexone, 200 mg/day of sertraline, and individual, cognitive behavioral therapy (CBT). For testing the medication, the design will be 2x2, consisting of four groups: naltrexone/sertraline, naltrexone only, sertraline only, placebo. All four groups will receive once weekly sessions of CBT given by therapists experienced in working with patients with substance disorders and trained in the principles of CBT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 75 years of age.
* Patients must have met DSM-IV criteria for (primary or substance-induced) major depressive episode prior to randomization.
* Patients must have a current DSM-IV diagnosis of alcohol dependence.
* Patients must have a total score of 10 or higher on the Hamilton Depression Scaleat the day of randomization. Also, item 1 on the scale must be > 1.
* Patients must have drank sufficient alcohol in the month prior to coming for treatment so that a practical assessment in reductions in drinking during and after treatment can be performed. The guidelines we will follow for this study as to what we think is sufficient will be that the patient in the month prior to coming to treatment will have drank on 40% or more of the days or drank more than 40 standard drinks (an average of 10 drinks per week).
* Patients must have successfully completed medical detoxification for alcohol (are abstinent for 4 consecutive days) or if medical detoxification is not indicated, have been abstinent for 4 consecutive days since coming to treatment but before initiating the study medication/placebo.
* Females of childbearing potential must have a negative pregnancy test and not contemplating pregnancy within the next 6 months. They must also use a contraceptive method judged by the investigator to be effective.

Exclusion Criteria:

* Patients with evidence of opiate use in the past 30 days as assessed by self-report and intake urine drug screens (only one repeat testing permitted). Patients with a history of treatment for opiate dependence will be excluded.
* Patients who, within the past year, met DSM IV criteria for dependence on any psychoactive substance other than alcohol or nicotine. Patients who test positive on the urine drug screen (with the exception of THC) at the initial visit (only one repeat testing permitted).
* Patients who meet DSM-IV criteria for past history or current disorder of schizophrenia or any psychotic disorder, or bipolar disorder.
* Patients with evidence or history of significant hematological, pulmonary, endocrine, cardiovascular, renal or gastrointestinal disease. (If there is a history of such disease but the condition has been stable for more than one year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.)
* Patients with abnormal liver function tests (AST or ALT) (more than 3.5 times the upper level of the normal value) or patients with any abnormal elevation in bilirubin.
* Patients requiring concomitant therapy with any psychotropic drug (with the exception of benadryl used sparingly if necessary for sleep or oxeazepam for detoxification or nicotine replacement therapy).
* Patients who have taken fluoxetine (Prozac) during the 6 weeks prior to randomization --due to its long half-life.
* Patients who have taken monoamine oxidase inhibitors (MAOI) during the 2 weeks prior to randomization -- due to the potential toxicity of combining MAOI medications with serotonin-specific ones. (Patients will also be instructed not to take MAOI for 2 weeks after completing the study.)
* Past use of antidepressants or other psychotropic medications (except as specified above) within 7 days of randomization.
* Patients on concomitant therapy with an investigational drug, or patients who have been in an investigational drug study within one month prior to entering this study.
* Patients who are unable to read or print in English.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2000-01; Primary Completion 2005-08 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Subjects self-report of alcohol use, measured by the Timeline Followback (TLFB), and depressive symptoms measured by scores on the Beck Depression Inventory (BDI) and Hamilton Rating Scale for Depression (HRSD). | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen Pettinati, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Treatment Research Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Pettinati HM, Oslin DW, Kampman KM, Dundon WD, Xie H, Gallis TL, Dackis CA, O'Brien CP. A double-blind, placebo-controlled trial combining sertraline and naltrexone for treating co-occurring depression and alcohol dependence. Am J Psychiatry. 2010 Jun;167(6):668-75. doi: 10.1176/appi.ajp.2009.08060852. Epub 2010 Mar 15. PMID 20231324